CLINICAL TRIAL: NCT04883099
Title: 7 Day Trial of APIOC for Presbyopia and APIOC for Presbyopia With Astigmatism
Brief Title: APIOC for Presbyopia and APIOC for Presbyopia With Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lentechs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEN101
Record Dates: First submitted 2021-05-04; First posted 2021-05-12 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Presbyopia; Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Presbyopia; Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- APIOC for Presbyopia and Presbyopia with Astigmatism (Experimental): Presbyopic Spherical or Toric Contact Lens
  Interventions: Device: APIOC for Presbyopia and APIOC for Presbyopia for Astigmatism

INTERVENTIONS:
Device: APIOC for Presbyopia and APIOC for Presbyopia for Astigmatism — Contact Lenses for Presbyopia

SUMMARY:
Vision and comfort, both objective and subjective, will be assessed for single vision contact lens wearers for either the APIOC™ for Presbyopia or the APIOC™ for Presbyopia Astigmatism contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must provide written informed consent.
2. The subject must appear willing and able to adhere to the instructions set forth in this protocol.
3. At least 40 years of age and no more than 70 years of age.
4. ≤ 4.00 D of corneal astigmatism.
5. ≤ 2.50 D of refractive astigmatism.
6. Refractive error range +4.00 DS to -6.00 DS
7. Require a reading addition (bifocal) of at least 0.75 D
8. Flat and steep keratometry readings within 40 to 48 D.
9. Clear, healthy corneas with no irregular astigmatism.
10. Normal, healthy conjunctiva in both eyes.
11. Free of active ocular disease. Refractive error and presbyopia are permitted.
12. Be a current or former (within the last 3 years) contact lens wearer.
13. Best-corrected near and distance visual acuity better than or equal to 20/25.

Exclusion Criteria:

1. Irregular corneal astigmatism.
2. Corneal scarring unless off line-of-site and well healed.
3. Pinguecula, pterygium, or other conjunctival thickness abnormalities that would interfere with soft contact lens wear.
4. Recent use of any ocular pharmaceutical treatments, including daily artificial tears, in the two weeks prior to the examination. Occasional artificial tear use is permitted.
5. Systemic disease that would interfere with contact lens wear.
6. Currently pregnant or lactating (by self-report).
7. History of strabismus or eye movement disorder, including exophoria at near that is 4 D or greater than at far, and a receded near point of convergence break that is 6 cm or greater.
8. Active allergies that may inhibit contact lens wear.
9. Upper eyelid margin at or above the superior limbus.
10. History of ocular or lid surgery.
11. Immediate family members or significant others of doctors or staff at the clinical site.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Visual Acuity Distance | Day 7
  High and Low Contrast LogMAR
Subjective Vision Quality | Day 7
  Visual analogue scale (0-100 points) 100 is best possible quality of vision
Comfort | Day 7
  Visual analogue scale(0-100 points) 100 is best possible comfort
Visual Acuity Near | Day 7
  High and Low Contrast
Visual Acuity Intermediate | Day 7
  High and Low Contrast

SECONDARY OUTCOMES:
Subjective Comfort | Day 7
  Compared to habitual lenses, rated as better/same/worse
Subjective vision Comparison | Day 7
  Compared to habitual lenses, rated as better/same/worse

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Quinn, OD, MS, Principal Investigator — Athens Eye Care
Locations (6):
- United States (6):
  - Complete Family Vision Care, San Diego, California
  - Eola Eyes, Orlando, Florida
  - Gaddie Eye Centers, Lexington, Kentucky
  - Miamisburg Vision Care, Miamisburg, Ohio
  - Vision Professionals, New Albany, Ohio
  - Eyecare Professionals of Powell, Powell, Ohio

IPD SHARING:
Plan to Share IPD: No
No sharing of data is planned.